CLINICAL TRIAL: NCT05201742
Title: A Comparative Study of Incentive Spirometer Versus Inspiratory Muscle Trainer on Pulmonary Function in Patients With Parkinsonism
Brief Title: Incentive Spirometer and Inspiratory Muscle Trainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GSITESC/24/16
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Incentive spirometer; Inspiratory muscle trainer; Pulmonary functions
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle trainer (Active Comparator): Inspiratory muscle trainer group - Inspiratory muscle training was performed.
  Interventions: Other: Inspiratory muscle training
- Incentive spirometer (Active Comparator): Incentive spirometer group - Incentive spirometry was performed.
  Interventions: Other: Incentive Spirometry

INTERVENTIONS:
Other: Inspiratory muscle training — Threshold inspiratory muscle training was performed for 6 weeks with device.
  Arms: Inspiratory muscle trainer
Other: Incentive Spirometry — Incentive spirometry was performed for 6 weeks with device.
  Arms: Incentive spirometer

SUMMARY:
Patients suffering from parkinsonism have respiratory function abnormalities. This study compared the effects of incentive spirometer and inspiratory muscle trainer on pulmonary functions in patients with parkinsonism.

DETAILED DESCRIPTION:
The participants were recruited according to the inclusion and exclusion criteria. Participants were divided into two groups - incentive spirometer and inspiratory muscle trainer. These trainings were performed for 6 weeks duration. Several outcome measures related to pulmonary function tests were measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having Parkinsonism Disease by the Neuro physician.
* Duration of Parkinson's Disease ≥ 5 years.
* Patients with the age of 65 to 80 years.
* Hoen and Yahr classification within 1 to 3.
* Both males and females were included.
* Patients who were able to comprehend the commands.
* Patients who were willing to participate.

Exclusion Criteria:

* Patients having any cardiovascular and pulmonary disorders.
* History of smoking currently or in the past.
* Psychological Impairment.
* Insufficient verbal/intellectual understanding.
* Patients with unstable vital parameters.
* Those unable to perform pulmonary function tests (PFT) because of anatomical abnormalities or clinical signs of dementia.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory pressure (MIP) | 6 weeks
  Maximum inspiratory pressure was measured.
6-minute walk distance (6 MWD) | 6 weeks
  Distance walked by the patients in 6 minutes was measured.
Forced vital capacity (FVC) | 6 weeks
  Forced vital capacity was measured.
Forced expiratory volume in 1 second (FEV1) | 6 weeks
  Forced expiratory volume in 1 second was measured
Peak Expiratory Flow Rate (PEFR) | 6 weeks
  Peak Expiratory Flow Rate was measured

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No